CLINICAL TRIAL: NCT03162198
Title: Frequency of Circulating Tumor Cells (CTCs) and Amount of Cell-free DNA (cfDNA) in Cirrhotic Patients With Hepatocellular Carcinoma (HCC)
Status: Completed | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-HCC-03
Record Dates: First submitted 2017-04-20; First posted 2017-05-22 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cirrhosis with HCC
  Interventions: Other: Cirrhosis with HCC
- Cirrhosis without HCC
  Interventions: Other: Cirrhosis without HCC

INTERVENTIONS:
Other: Cirrhosis with HCC — Cirrhosis with Hepatocellular Carcinoma
  Groups: Cirrhosis with HCC
Other: Cirrhosis without HCC — Cirrhosis without Hepatocellular Carcinoma
  Groups: Cirrhosis without HCC

SUMMARY:
All consecutive patients with liver cirrhosis, with clinical and imaging features suggestive of Hepatocellular Carcinoma (HCC) attending the Department of Hepatology, Institute of Liver and Biliary Sciences (ILBS) from February 2017 to December 2018 will be evaluated for inclusion.Based on the previous years data of HCC patients admitted to ILBS.

Cirrhotic patients aged 18-70 years, with HCC proven by typical radiological features of arterial enhancement and delayed wash-out, on one or both of dynamic Computerized Tomographic or dynamic Magnetic Resonance Imaging (MRI), as per updated American Association for the Study of Liver Disease (AASLD) guidelines (details in appendix1).

Age and gender matched patients with cirrhosis, but without HCC, seen during the same study period will serve as controls.

Patient characteristics, etiology of cirrhosis, and liver function parameters will be noted. Investigator will stage the included patients as per the Barcelona Cancer of Liver Cancer (BCLC) criteria (details in appendix1). Investigator will then estimate Circulating Tumor Cells (CTC) and cfDNA in peripheral blood samples of the patients and controls.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-70 years.
* Proven cirrhosis (Defined in appendix 1).
* HCC proven by standard radiological criteria within last 1-month (For Cases)
* No HCC on dynamic CT and/or dynamic MRI (protocol defined in appendix 1) done within last 1 month (For Control Group).

Exclusion Criteria:

* Previous biopsy or FNA of the tumor.
* Previous invasive radiological procedures TACE/RFA.
* Previous or ongoing chemotherapy or biological therapy.
* Previous liver resection or transplant.
* Segmental / main PV thrombosis.
* Atypical enhancement on imaging
* Extrahepatic metastatic spread of HCC
* >70 years of age
* Coexisting sepsis.
* Renal dysfunction, as defined by serum creatinine >1.5mg/dL.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Proven cirrhosis with HCC proven by standard radiological criteria within last 1 month.
  * Proven cirrhosis with no HCC on dynamic CT and/or dynamic MRI done within last 1 month.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Number of circulating tumor cells (CTCs) in cirrhotic patients with hepatocellular carcinoma (HCC) | Day 0
Number of cell-free DNA (cfDNA) in cirrhotic patients with hepatocellular carcinoma (HCC) | Day 0

SECONDARY OUTCOMES:
Number of Circulating Tumor Cells in the peripheral blood of cirrhotic patients in both groups | Day 0
To study the difference in amount of cfDNA in the peripheral blood of cirrhotic patients with and without HCC. | Day 0
  Difference would be found out by estimating cfDNA in terms of ng/mL of the blood specimen
Number of Circulatory Tumor Cells with the tumor size of HepatoCellular Carcinoma. | Day 0
Number of Circulatory Tumor Cells with the tumor number of HepatoCellular Carcinoma. | Day 0
Number of Circulatory Tumor Cells withBarcelona Clinic of Liver Cancer (BCLC) stage of HepatoCellular Carcinoma. | Day 0
Number of cfDNA amount with the tumor size of HepatoCellular Carcinoma. | Day 0
Number of cfDNA amount with the tumor number of HepatoCellular Carcinoma. | Day 0
Number of cfDNA amount with the Barcelona Clinic of Liver Cancer (BCLC) stage of HepatoCellular Carcinoma. | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No